CLINICAL TRIAL: NCT04805034
Title: Predictive Model for Prognosis of E Antigen-positive Mothers With Chronic HBV Infection: A Multicenter Cohort Study
Brief Title: Predictive Model for Prognosis of Chronic HBV Infection Mothers
Acronym: PMFPOEPMWCHI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: the Second Affiliated Hospital of Shaanxi University of Traditional Chinese Medicine (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Shaanxi Provincial People's Hospital (Other); Baoji Maternal and Child Health Hospital (Unknown); Weinan Central Hospital (Other); Ankang Central Hospital (Other); Hanzhong Central Hospital (Other); Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2020-001
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBeAg positive/HBsAg positive
  Interventions: Other: Age, BMI,Baseline HBV DNA, Baseline HBeAg level, Baseline HBsAg level, Antiviral treatment, Serum ALT level
- HBeAg seroconversion /HBsAg loss
  Interventions: Other: Age, BMI,Baseline HBV DNA, Baseline HBeAg level, Baseline HBsAg level, Antiviral treatment, Serum ALT level

INTERVENTIONS:
Other: Age, BMI,Baseline HBV DNA, Baseline HBeAg level, Baseline HBsAg level, Antiviral treatment, Serum ALT level — Exposure factors: Age, BMI, Family history, Baseline HBV DNA, Baseline HBeAg level, Baseline HBsAg level, Antiviral treatment, Serum ALT level

SUMMARY:
Pregnancy is a complex and coordinated physiological process. Pregnancy and the postpartum period are associated with unique changes in the immune system that may impact the natural history of autoimmune diseases and immune-mediated infections. In the postpartum period. ALT ﬂares have been reported in 20%-60% of untreated women and were more likely to occur in hepatitis B e antigen (HBeAg)-positive patients. It has been postulated that postpartum ALT ﬂares may arise to rapid immune restitution against hepatitis B virus (HBV) antigens in the liver, when may be a timing of antiviral treatment. A large number of previous studies have focused on studies on the interruption of mother-to-child transmission in women with chronic hepatitis B(CHB), but studies on the prognosis of mothers undergoing pregnancy and delivery are very limited. What are the factors that affect the clearance of HBeAg or HBsAg? What kind of antiviral treatment protocol should be adopted for mothers with CHB? It is not only a problem that needs to be solved urgently in clinical practice, but also can provide some clues for understanding the occurrence and development of HBV infection in women of childbearing age.

Overall, this study intends to carry out a multi-center two-way cohort study on E antigen-positive CHB women in 9 hospitals in Shaanxi Province. To observe the dynamic changes of virological parameters in these patients, figure out the factors of the serum HBsAg loss and HBeAg seroconversion, and establish relevant predictive models.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-45 years old
* Serum HBsAg positive> 6 months
* HBeAg positive at delivery
* Good compliance

Exclusion Criteria:

* Women who give birth to stillbirth due to various reasons
* Coinfection with HIV,HCV, syphilis or other sexually transmitted diseases
* Severe kidney, cardiovascular, lung, nervous system or immune system diseases
* Who are taking immunotherapy drugs or anti-tumor drugs

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mothers with chronic hepatitis B infection
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
the rate of HBeAg loss | Postpartum 96weeks
the rate of HBeAg seroconversion | Postpartum 96weeks
the rate of HBsAg loss | Postpartum 96weeks

SECONDARY OUTCOMES:
the rate of undetectable HBV DNA | Postpartum 96weeks
the rate ALT normalization | Postpartum 96weeks
Dynamic changes of serum HBsAg, HBeAg, HBV DNA and HBV RNA titer | at delivery, 12 weeks, 24 weeks, 48 weeks, 72 weeks, 96 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tianyan Chen, phD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided